CLINICAL TRIAL: NCT05575856
Title: Cardiogenic Shock Registry Mannheim - CARESMA
Brief Title: Cardiogenic Shock Registry Mannheim
Acronym: CARESMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Prof. Dr., Universitätsmedizin Mannheim
Other Study IDs: 2019-695N
Record Dates: First submitted 2022-03-12; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock; heart failure; cardiac arrest; shock; acute myocardial infarction
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure; Heart Arrest; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to investigate clinically and prognostically relevant parameters in patients with cardiogenic shock within a monocentric observational clinical register.

DETAILED DESCRIPTION:
All consecutive patients with a confirmed cardiogenic shock presenting at the internal intensive care Unit (ICU) at the University of Mannheim are included in the register and followed up during ICU stay and after that. Data of patients' admission status, cause of cardiogenic shock, baseline parameters and comorbidities are collected. Extensive information about echocardiography, electrocardiography and imaging procedures are included in the register. Laboratory values, microbiological investigations, organ dysfunction and organ replacement therapies, medication, adverse events, and complications were recorded for several days during the ICU stay (days 1, 2, 3, 5, 7, and 8). Standard scores for critically ill patients were calculated for the day of admission at the ICU if available, and several time points during the ICU stay. The register includes information about the mortality during ICU stay, 30-day mortality, 6-month mortality and 1-year mortality.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock according to current guidelines

Exclusion Criteria:

* other forms of shock not primary associated with cardiac dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all patients presenting with a cardiogenic shock at the intensive care unit (ICU).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 30 days
  days

SECONDARY OUTCOMES:
all-cause mortality | during hospital stay (up to 30 days)
  during hospital stay (up to 30 days)
all-cause mortality | 1 years
  years
ventilator-free days | 30 days
  days

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Medicine, University Medical Centre Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rusnak J, Schupp T, Weidner K, Ruka M, Egner-Walter S, Schmitt A, Akin M, Tajti P, Mashayekhi K, Ayoub M, Behnes M, Akin I. Prognostic Influence of Lung Compliance in Patients with Cardiogenic Shock and Invasive Mechanical Ventilation. Rev Cardiovasc Med. 2024 Nov 22;25(11):420. doi: 10.31083/j.rcm2511420. eCollection 2024 Nov. PMID 39618866
- [Derived] Rusnak J, Schupp T, Weidner K, Ruka M, Egner-Walter S, Forner J, Schmitt A, Akin M, Tajti P, Mashayekhi K, Ayoub M, Akin I, Behnes M. Influence of Right and Left Bundle Branch Block in Patients With Cardiogenic Shock and Cardiac Arrest. Crit Care Med. 2025 Jan 1;53(1):e54-e64. doi: 10.1097/CCM.0000000000006459. Epub 2024 Oct 29. PMID 39470337
- [Derived] Schupp T, Rusnak J, Forner J, Dudda J, Bertsch T, Behnes M, Akin I. Platelet Count During Course of Cardiogenic Shock. ASAIO J. 2024 Jan 1;70(1):44-52. doi: 10.1097/MAT.0000000000002066. Epub 2023 Oct 12. PMID 37831815
- [Derived] Behnes M, Rusnak J, Egner-Walter S, Ruka M, Dudda J, Schmitt A, Forner J, Mashayekhi K, Tajti P, Ayoub M, Weiss C, Akin I, Schupp T. Effect of Admission and Onset Time on the Prognosis of Patients With Cardiogenic Shock. Chest. 2024 Jan;165(1):110-127. doi: 10.1016/j.chest.2023.08.011. Epub 2023 Aug 12. PMID 37579943
- [Derived] Schmitt A, Schupp T, Rusnak J, Ruka M, Egner-Walter S, Mashayekhi K, Tajti P, Ayoub M, Behnes M, Akin I, Weidner K. Does sex affect the risk of 30-day all-cause mortality in cardiogenic shock? Int J Cardiol. 2023 Jun 15;381:105-111. doi: 10.1016/j.ijcard.2023.03.061. Epub 2023 Mar 31. PMID 37004944